CLINICAL TRIAL: NCT05406713
Title: Neoadjuvant Pembrolizumab in Patients With Muscle-invasive Bladder Cancer With Selective Bladder Sparing
Brief Title: Pembrolizumab in Muscle-invasive Bladder Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew Galsky (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Matthew Galsky, Principal Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU20-444
Record Dates: First submitted 2022-05-09; First posted 2022-06-06 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Muscle Invasive Bladder Carcinoma; Localized Cancer; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Group (Experimental): Cycles 1-2 (Pembrolizumab): 400 mg of Pembrolizumab intravenously (Administered Day 1 of 42 day Cycle)
  If complete response of treatment is observed then maintenance therapy will be given. All other patients will receive with standard of care local therapy (cystectomy or chemo-radiation) as per their treating physicians followed by "adjuvant" pembrolizumab.
  Cycle 3-9 (Maintenance or Adjuvant Single agent Pembrolizumab): 400 mg of Pembrolizumab intravenously (Administered Day 1 of 42 day Cycle)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 400 mg intravenously
  Other Names: Keytruda

SUMMARY:
Subjects with cT2-T3N0M0 urothelial cancer of the bladder will be enrolled. After completing two cycles of pembrolizumab, subjects will undergo a restaging MRI of the abdomen and pelvis with a standard acquisition protocol (as outlined in the protocol) as well as CT chest. A CT of the abdomen and pelvis may be performed if there are contraindications to MRI. Patients will also undergo a restaging cystoscopy and biopsies/TURBT as outlined in the protocol.

Patients achieving a clinical complete response to treatment (defined in the protocol) will proceed with "maintenance" single agent pembrolizumab followed by surveillance. All other patients will proceed with standard of care local therapy as per their treating physicians followed by "adjuvant" pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of ≤ 1 within 28 days prior to registration.
* Histological evidence of clinically localized muscle-invasive urothelial cancer of the bladder. Clinical stage cT2-3N0M0. N0 will be considered the absence of radiographically enlarged lymph nodes on baseline imaging. Patients with lymph nodes <1 cm in long axis on imaging may be eligible but must be discussed with the sponsor investigator.
* Have undergone a standard of care maximal transurethral resection of bladder tumor ≤ 60 days prior C1D1. Maximal TURBT is defined as a macroscopically complete resection of bladder tumor when safely possibly per the treating urologist. Patients who cannot safely undergo maximal TURBT as per their treating urologist are eligible for enrollment but should be discussed with the sponsor investigator.
* All subjects must have adequate transurethral resection of bladder tumor tissue available for submission (i.e., at least 15 unstained slides or paraffin block) identified during screening. This tissue can be from the maximal restaging TURBT, a prior diagnostic TURBT revealing muscle-invasive bladder cancer, or both specimens. Subjects without available archival tissue must be discussed with the sponsor-investigator.
* Decline cisplatin-based neoadjuvant chemotherapy or be considered cisplatin-ineligible based on at least one of the following modified criteria (as ECOG 0-1 is required for eligibility):

  * Creatinine clearance < 60 mL/min (but ≥ 30 mL/min)
  * Grade ≥ 2 hearing loss (per CTCAE criteria v5)
  * Grade ≥ 2 neuropathy (per CTCAE criteria v5)
  * New York Heart Association Class III heart failure
* Demonstrate adequate organ function as defined below. All screening labs to be obtained within 28 days prior to registration.

  * Hematological

    * Absolute Neutrophil Count (ANC): ≥ 1.5 x 10^9/L
    * Hemoglobin (Hgb): ≥ 9 g/dL
    * Platelets: ≥ 100 x 10^9/L
  * Renal

    * Creatinine OR: Creatinine ≤ 1.5 × ULN OR
    * Calculated creatinine clearance: creatinine clearance ≥ 30 mL/min
  * Hepatic

    * Bilirubin: ≤ 1.5 ×ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN
    * Aspartate aminotransferase (AST): ≤ 2.5 × ULN
    * Alanine aminotransferase (ALT): ≤ 2.5 × ULN
* Women of childbearing potential (WOCP) must have a negative serum or urine pregnancy test a maximum of 24-hours before the first dose of study drug. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. WOCBP must agree to use contraception.
* A male participant must agree to use contraception.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Prior systemic chemotherapy for muscle-invasive urothelial cancer of the bladder.
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured. Patients with intermediate or lower risk prostate cancer as defined by the National Comprehensive Cancer Network (NCCN) risk stratification guidelines may be eligible for enrollment.
* Prior radiation therapy for bladder cancer.
* Active infection requiring systemic therapy.
* Has a known history of Hepatitis B or C. NOTE: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. NOTE: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a known history of Human Immunodeficiency Virus (HIV) infection. NOTE: no testing for HIV is required unless mandated by local health authority.
* Has a known history of active TB (Bacillus Tuberculosis).
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has had an allogenic tissue/solid organ transplant.
* Is currently receiving an investigational agent or has received an investigational agent or used an investigational device within 28 days of study registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Complete Response Rate (CRR) | 2 years
  Estimate the clinical complete response rate defined as cT0 or cTa disease after pembrolizumab
Benefit from Treatment | 2 years
  Estimate the ability of clinical complete response (cT0 or cTa) to predict benefit from treatment. For patients achieving a clinical complete response, benefit will be defined as 2 year metastasis-free survival in patients among the patients achieving a clinical complete response.

SECONDARY OUTCOMES:
Assess adverse events | 6 months
  Describe the safety of neoadjuvant pembrolizumab.Safety will be determined according to the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v5
Positive Predictive Value between PD-L1 Expression and clinical complete response | 2 years
  Positive predictive value of PD-L1 CPS, in predicting benefit from treatment in patients achieving a clinical complete response. Combined Positive Score (CPS) is defined as the number of PD-L1 staining cells divided by the total number of viable tumor cells, multiplied by 100.
Positive Predictive Value between TMB and clinical complete response | 2 years
  Positive predictive value of TMB in predicting benefit from treatment in patients achieving a clinical complete response. Tumor mutational burden (TMB) is defined as the total number of somatic nonsynonymous mutations per coding area of a tumor genome.
Metastasis Free Survival | 2 years
  Estimate metastasis free survival in the overall study population. Metastasis-free survival is defined as the time from initiation of treatment to the development of metastatic disease. Microscopic metastatic disease involving regional lymph nodes resected at cystectomy performed with curative intent will not be considered an event. Confirmation of metastatic recurrence with a biopsy is recommended in all situations.
Metastasis Free Survival | 2 years
  Estimate the 2 year metastasis-free survival. Metastasis-free survival is defined as the time from initiation of treatment to the development of metastatic disease. Microscopic metastatic disease involving regional lymph nodes resected at cystectomy performed with curative intent will not be considered an event. Confirmation of metastatic recurrence with a biopsy is recommended in all situations.
Metastasis Free Survival | 2 years
  Estimate metastasis free survival in patients achieving a clinical complete response. Metastasis-free survival is defined as the time from initiation of treatment to the development of metastatic disease. Microscopic metastatic disease involving regional lymph nodes resected at cystectomy performed with curative intent will not be considered an event. Confirmation of metastatic recurrence with a biopsy is recommended in all situations.
Metastasis Free Survival | 2 years
  Estimate metastasis free survival in patients not achieving a clinical complete response. Metastasis-free survival is defined as the time from initiation of treatment to the development of metastatic disease. Microscopic metastatic disease involving regional lymph nodes resected at cystectomy performed with curative intent will not be considered an event. Confirmation of metastatic recurrence with a biopsy is recommended in all situations.
Bladder-intact Event Free Survival | 2 years
  Bladder-intact event-free survival is defined from initiation of treatment until radical cystectomy, evidence of unresectable or metastatic disease, or death due to any cause.
Bladder-intact Event Free Survival | 2 years
  Estimate bladder-intact event free survival in patients achieving a clinical complete response. Bladder-intact event-free survival is defined from initiation of treatment until radical cystectomy, evidence of unresectable or metastatic disease, or death due to any cause.
Bladder-intact Event Free Survival | 2 years
  Estimate bladder-intact event free survival in patients not achieving a clinical complete response. Bladder-intact event-free survival is defined from initiation of treatment until radical cystectomy, evidence of unresectable or metastatic disease, or death due to any cause.
Overall Survival (OS) | 2 years
  Estimate overall survival. Overall survival is defined as the time from initiation of treatment to death.
Overall Survival (OS) | 2 years
  Estimate overall survival in patients achieving a clinical complete response. Overall survival is defined as the time from initiation of treatment to death.
Overall Survival (OS) | 2 years
  Estimate overall survival in patients not achieving a clinical complete response. Overall survival is defined as the time from initiation of treatment to death.
Bladder-Intact Overall Survival | 2 years
  Estimate bladder-intact overall survival. Bladder-intact overall survival is defined as the time from initiation of treatment until death or cystectomy.
Bladder-Intact Overall Survival | 2 years
  Estimate bladder-intact overall survival in patients achieving a clinical complete response. Bladder-intact overall survival is defined as the time from initiation of treatment until death or cystectomy.
Bladder-Intact Overall Survival | 2 years
  Estimate bladder-intact overall survival in patients not achieving a clinical complete response. Bladder-intact overall survival is defined as the time from initiation of treatment until death or cystectomy.
Invasive Bladder Recurrence Free Survival | 2 years
  Estimate invasive bladder recurrence-free survival in patients achieving a clinical complete response and in all patients not undergoing cystectomy. Invasive bladder recurrence free survival will be defined as the time from initiation of treatment to the development of at least cT/pT1 urothelial cancer in the bladder.
Recurrence Free Survival (RFS) | 2 years
  Estimate the RFS. Recurrence-free survival is defined as the time from initiation of treatment to death or recurrence, depending on which occurs first.
Recurrence Free Survival (RFS) | 2 years
  Estimate the RFS in patients achieving a clinical complete response. Recurrence-free survival is defined as the time from initiation of treatment to death or recurrence, depending on which occurs first.
Recurrence Free Survival (RFS) | 2 years
  Estimate the RFS in patients not achieving a clinical complete response. Recurrence-free survival is defined as the time from initiation of treatment to death or recurrence, depending on which occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Galsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - City of Hope, Duarte, California
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No